CLINICAL TRIAL: NCT01111422
Title: A Randomized Prospective Trial of N-acetyl Cystein in Patients With Peritoneal Dialysis
Brief Title: Anti-Oxidant Effect on Peritoneal Membrane in Peritoneal Dialysis (PD) Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University (Other)
Responsible Party: Nephrology, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ewha 219-3-40
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-03

CONDITIONS: End-Stage Kidney Disease; Peritoneal Dialysis
Keywords: Antioxidant; Epithelial to Mesenchymal Transition; peritoneal fibrosis; Peritoneal Dialysis, Continuous Ambulatory
MeSH Terms: conditions — Kidney Failure, Chronic; Peritoneal Fibrosis | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Age and sex matched peritoneal dialysis patients
- N-acetylcysteine (Experimental): N-acetylcysteine in stable peritoneal dialysis patients
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine (200 mg/capsule) 1200 mg/day (600 mg bid) for 6 months
  Other Names: Muteran capsuleⓇ HAN WHA PHARM.
  Arms: N-acetylcysteine

SUMMARY:
Peritoneal fibrosis is one of the major causes of technical failure in patients on peritoneal dialysis (PD) for long period of time. Although the exact mechanisms of peritoneal damage during PD still remain unclear, generation of reactive oxygen species may be responsible for progressive membrane dysfunction. N-acetylcysteine (NAC)is a powerful antioxidant shown to protect peritoneal fibrosis in peritoneal dialysis animal model. In this study the researchers investigated the hypothesis that NAC protect peritoneal membrane damage.

DETAILED DESCRIPTION:
N-Acetylcysteine (NAC) is known to be relatively safe and beneficial in peritoneal dialysis patient at a dose of 1200 mg per day. Patients will be randomly assigned to NAC and control group and prescribed according to the protocol. At 2 and 6 month, Peritoneal equilibrium test (PET) will be performed with blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance peritoneal dialysis at least 3 months
* Patients who are able and willing to understand, sign and date an informed consent document, and authorize access to protected health information

Exclusion Criteria:

* Episode of peritonitis at least 3 months
* Episodes of admission due to other disease at lease 3 months
* Liver disease
* Allergic history with N-acetylcysteine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Peritoneal membrane function | 6 months
  Changes in peritoneal membrane function (Δ D/Pcreatinine, ΔD/Purea) with peritoneal equilibrium test

SECONDARY OUTCOMES:
Oxydative stress status | 6 months
  Measurement of oxydative stress status with plasma and RBC (GSH/GSSG, 8-OHdG)
Mesothelial cell transformation (Epithelial to Mesenchymal Transition) | 6 month
  Morphology was analysed with peritoneal dialysate isolated mesothelial cell
Residual renal function | 6 month
  Changes in residual renal function (ΔKt/Vurea, ΔeGFR)
Peritoneal membrane function | 2 months
  Changes in peritoneal membrane function (Δ D/Pcreatinine, ΔD/Purea) with peritoneal equilibrium test

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hee Kang, MD. PhD., Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea